CLINICAL TRIAL: NCT05273892
Title: King's Intervention to Achieve Nutrition & Exercise Goals Supported by Lifestyle Advice for Desk-based/Work From Home Workers Delivered as a HOListic Employee Wellbeing Programme: The KING'S WHOLE Feasibility Study
Brief Title: The KING'S WHOLE Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KT 2021
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-03

CONDITIONS: Overweight or Obesity
Keywords: Employee; Lifestyle intervention; Online health and wellbeing
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet; Exercise; Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet + Activity + Sleep (Experimental)
  Interventions: Behavioral: Diet + Activity + Sleep
- Diet + Activity (Active Comparator)
  Interventions: Behavioral: Diet + Activity

INTERVENTIONS:
Behavioral: Diet + Activity + Sleep — Personalized lifestyle behavior change counselling
  Arms: Diet + Activity + Sleep
Behavioral: Diet + Activity — Personalized lifestyle behavior change counselling
  Arms: Diet + Activity

SUMMARY:
Office working life has changed dramatically over the last 50 years with digitalization; this is estimated to have decreased the amount of energy (calories) used during work. Employees who work long or irregular working hours or experience job strain are more likely to make less healthy food choices. The combination of these factors may contribute to increased body weight during a persons working life. The aim is to investigate the feasibility of an online lifestyle behaviour change intervention in office workers.

DETAILED DESCRIPTION:
Office working life has changed dramatically over the last 50 years with digitalization; this is estimated to have decreased the amount of energy (calories) used during work. Employees who work long or irregular working hours or experience job strain are more likely to make less healthy food choices. The combination of these factors may contribute to increased body weight during a persons working life. The aim is to investigate the feasibility of an online lifestyle behaviour change intervention in office workers.

This feasibility randomized control trial is a remote study and will be conducted online. Participants will be randomized to one of two health and well being interventions.

The study will last 14 weeks. Participants need to attend two on-line study appointments (at the start of week 1 and end of week 14) lasting approximately 30-45 minutes.

In weeks 2, 6 and 10 participants will be asked to participate in a personalised one-to-one behaviour change on-line advice session with a research nutritionist/dietitian. Each session will last approximately 45 minutes.

In weeks 1, 5, 9 and 14 participants will be asked to wear a wrist-worn activity monitor and report what you eat and drink for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* King's College employee (working at least 0.5 WTE)
* Work in a desk/computer-based job role
* Body mass index (BMI) that is more than 25kg/m2 and waist circumference indicative of increased cardiometabolic risk based on NHS guidelines for different ethnic groups by sex: Men - White waist circumference more than 94cm (37-in); men of Chinese, Asian, African or African-Caribbean ethnicity - more than 90cm (35.4in). Women - waist circumference more than 80 cm (31.5in)
* Sleep duration 5 - <7 hours on average on most weekdays
* Not actively loosing weight or part of weight management programme (e.g., Weight Watchers or Slimming World)
* Not under medical advice that contraindicates increasing physical activity and exercising.
* Not diagnosed with a sleep condition and have no history of chronic use of sleeping aids.
* Not diagnosed with an eating disorder.
* Not diagnosis in the last 12 months or currently requiring treatment for: heart attack, stroke, pacemaker, hepatitis or any liver disease, diabetes mellitus, chronic gastrointestinal disorders, thyroid conditions, or cancer (excluding basal carcinoma).
* No history of alcohol or drug misuse in the last 2 years.
* Own a smart phone and technology literate

Exclusion Criteria:

* - Shift worker (required to work outside 6 am and 8 pm)
* Pregnant / breastfeeding or have caring responsibilities that would prevent a participant from changing your daily routine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Engagement | 14 weeks
  Percentage of eligible volunteers consented
Attrition | 14 weeks
  Percentage drop out
Intervention adherence | 14 weeks
  Participants complying with intervention.
Intervention adherence - sleep | 14 weeks
  Sleep hygiene adherence; Scores will range from 0 - 52, with higher scores representing poorer sleep hygiene

SECONDARY OUTCOMES:
Change in body weight | 14 weeks
  Difference from baseline to post intervention in body weight (kg)
Change in energy and macro nutrient intake | 14 weeks
  Difference in energy intake (Kcal), and sources of energy (carbohydrates, fats, and protein)
Change in sleep duration | 14 weeks
  Difference in between baseline and post intervention (hours/night)
Change in physical activity intensity and duration | 14 weeks
  Difference in activity from MotionWatch (duration hours in vigorous and moderate activity)
Change in sleep quality score | 14 Weeks
  Difference in score from PROMIS (Patient-Reported Outcomes Measurement Information System) questionnaire. Scores between 8 and 40, which are converted to T-Scores (min 28.9 - 76.5). Higher score = more disturbance
Change in work engagement score | 14 Weeks
  Change in Utrecht Work Engagement Scale (UWES) questionnaire score. Three subscales for "Vigor", "dedication" "absorption" - all have score between 0 and 6. Higher scores = more vigor/dedication/absorption at work. 1 total UWEZ-9 Score. Score between 0 and 6. Higher score = more work engagement.
Change in anxiety questionnaire score | 14 weeks
  Difference in generalized anxiety (GAD-7) questionnaire score.Range 0 to 21. Higher score = higher anxiety level.
Change in depression questionnaire score | 14 weeks
  Difference in PHQ9 depression questionnaire score.Range 0 to 27. Higher score = more likely depressive symptoms.
Change in reported level of burn out | 14 weeks
  Difference in Oldenberg Burnout Inventory score, higher score = more burnout signs/symptoms
Change in day time sleepiness | 14 weeks
  Difference in Epworth Sleepiness Scale. Range 0 to 24 - higher score = more daytime sleepiness

OTHER OUTCOMES:
Change in job satisfaction score | 14 weeks
  Difference in job satisfaction questionnaire score.Score between 5 and 25. Higher score= more job satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Life Course Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided